CLINICAL TRIAL: NCT02240992
Title: Mesenchymal Stem Cells With or Without G-CSF Mobilized Peripheral Blood Stem Cell for Treatment of Poor Graft Function and Delayed Platelet Engraftment After Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: MSCs With or Without Peripheral Blood Stem Cell for Treatment of Poor Graft Function and Delayed Platelet Engraftment
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Guangzhou First People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Southern Medical University, China (Other); Peking University People's Hospital (Other); Huazhong University of Science and Technology (Other); Sun Yat-sen University (Other); Academy Military Medical Science, China (Industry)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFH-PBSC-MSC-PGF-2014
Record Dates: First submitted 2014-09-13; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Stem Cell Transplantation, Hematopoietic; Poor Graft Function; Delayed Platelet Engraftment; Hematological Diseases
Keywords: Poor Graft Function; Delayed platelet engraftment; Peripheral Blood Stem Cell; Mesenchymal Stem Cells; Allogeneic hematopoietic stem cell transplantation
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSCs&PBSC (Experimental): PBSC will be intravenously infused at a dose of 2×10^8/kg. MSCs will be intravenously infused at a dose of 1×10^6 cells/kg once per week or until complete response(CR) . If the patients do not achieve CR or partial remission (PR) within 4 weeks, they will swithed to other therapy. If the patients achieve PR within 4 weeks, a second course of the same treatment will be given.
  Interventions: Biological: PBSC; Biological: MSCs
- MSCs (Experimental): MSCs will be intravenously infused at a dose of 1×10^6 cells/kg once per week or until CR. If the patients have no response (NR) within 4 weeks, they will switch to other therapy. If the patients achieve PR within 4 weeks, a second course of the same treatment will be given.
  Interventions: Biological: MSCs

INTERVENTIONS:
Biological: PBSC
  Arms: MSCs&PBSC
Biological: MSCs

SUMMARY:
The purpose of this study is to compare the efficacy of mesenchymal stem cells (MSCs) with or without granulocyte colony-stimulating factor (G-CSF) mobilized peripheral stem cells (PBSC) in treating patients experiencing poor graft function or delayed platelet engraftment after allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation(allo-HSCT) is the only cure for many hematologic diseases. However, about 5-27% of patients would suffer from poor graft function (PGF) and more recipients might develop delayed platelet engraftment (DPE) after allo-HSCT. These complications are associated with considerable mortality related to infections or hemorrhagic complications. Treatment of PGF and DPE usually involves hematopoietic growth factors such as granulocyte colony-stimulating factor (G-CSF) and thrombopoietin (TPO), or second transplantation, but these methods have dismal effect or even a significant risk of graft-versus-host disease (GVHD).

Mesenchymal stem cells (MSCs) are a form of multipotent adult stem cells that can be isolated from bone marrow (BM), adipose tissue, and cord blood. Clinical applications of human MSCs include improving hematopoietic engraftment, preventing and treating graft-versus-host disease after allo-HSCT and so on. Some studies have shown that MSCs combined with PBSC or cord blood could be useful to improve engraftment after HSCT. Several reports suggested MSCs might be effective in the treatment of PGF.

However, the efficacy of MSCs as single-drug treatment for PGF or DPE is unsatisfactory in our previous study. Therefore, in the present study, G-CSF mobilized PBSC will be used combined with MSCs in the patients with PGF or DPE after allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Age：14-65 years
* PGF or DPE after allo-HSCT
* Subjects (or their legally acceptable representatives) must have signed an informed consent document

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Hematopoietic Recovery | 1 year
  Hematopoietic reconstitution post-transplantation is defined as reconstitution of both neutrophil and platelet numbers. Neutrophil reconstitution is defined as occurring on the first 3 consecutive days with an neutrophil(NEU)>0.5×10^9/L, and platelet (PLT) reconstitution is defined as the first >20×10^9/L for 3 consecutive days.

SECONDARY OUTCOMES:
Incidence of graft-versus-host disease | 1 year
  Graft-versus-host disease (GVHD) includes acute GVHD and chronic GVHD.
Incidence of infections | 1 year
  Infections include bacterial, invasive fungal and viral infections
Incidence of primary underlying disease relapse | 1 year
Incidence of acute toxicity | up to 100 days
  Acute toxicity mainly involves the heart,live and kidney.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Sanchez-Guijo FM, Lopez-Villar O, Lopez-Anglada L, Villaron EM, Muntion S, Diez-Campelo M, Perez-Simon JA, San Miguel JF, Caballero D, del Canizo MC. Allogeneic mesenchymal stem cell therapy for refractory cytopenias after hematopoietic stem cell transplantation. Transfusion. 2012 May;52(5):1086-91. doi: 10.1111/j.1537-2995.2011.03400.x. Epub 2011 Oct 24. PMID 22023454
- [Background] Meuleman N, Tondreau T, Ahmad I, Kwan J, Crokaert F, Delforge A, Dorval C, Martiat P, Lewalle P, Lagneaux L, Bron D. Infusion of mesenchymal stromal cells can aid hematopoietic recovery following allogeneic hematopoietic stem cell myeloablative transplant: a pilot study. Stem Cells Dev. 2009 Nov;18(9):1247-52. doi: 10.1089/scd.2009.0029. PMID 19309241